CLINICAL TRIAL: NCT06184425
Title: A Randomized Comparative Study Between 25-Gauge and 27-Gauage Pencil Point Spinal Needles During Dural Puncture Epidural Anaesthesia For Elective Caesarean Section
Brief Title: Dural Puncture Epidural Technique During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IF-2023
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia, Obstetric

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural Puncture Epidural technique using pencil-point 25G Whitacre needle (Active Comparator)
  Interventions: Procedure: Dural Puncture Epidural technique using pencil-point 27G Whitacre needle
- Dural Puncture Epidural technique using 27 G Whitacre needle (Experimental)
  Interventions: Procedure: Dural Puncture Epidural technique using pencil-point 25G Whitacre needle

INTERVENTIONS:
Procedure: Dural Puncture Epidural technique using pencil-point 25G Whitacre needle — - DPE technique was performed in the sitting position at the L3/4 or L4/5 interspace via the midline approach using a 17-gauge Touhy needle and a loss of resistance to saline technique, then the dura was punctured with a 25-gauge pencil point Whitacre spinal needles using a needle-through-needle technique, and spontaneous flow of cerebrospinal fluid was confirmed, then the spinal needle was removed and a flexible 19-gauge, spring closed-tip catheter was inserted 5 cm into the epidural space toward the cranial side.
  Arms: Dural Puncture Epidural technique using 27 G Whitacre needle
Procedure: Dural Puncture Epidural technique using pencil-point 27G Whitacre needle — - DPE technique was performed in the sitting position at the L3/4 or L4/5 interspace via the midline approach using a 17-gauge Touhy needle and a loss of resistance to saline technique, then the dura was punctured with a 27-gauage pencil point Whitacre spinal needles using a needle-through-needle technique, and spontaneous flow of cerebrospinal fluid was confirmed, then the spinal needle was removed and a flexible 19-gauge, spring closed-tip catheter was inserted 5 cm into the epidural space toward the cranial side.
  Arms: Dural Puncture Epidural technique using pencil-point 25G Whitacre needle

SUMMARY:
DPE technique was performed by creating a perforation in the dura mater using a pencil point spinal needle (25-27G) through the shaft of an epidural needle. After the dural perforation was created and the free flow of the cerebrospinal fluid (CSF) was confirmed, which was considered a definitive end point for the likely positioning of the epidural needle tip within the epidural space, and by avoiding direct intrathecal administration of medication making DPE technique of fewer adverse effects in comparison to CSE technique, then spinal needle was withdrawn without local anesthetic injection into the subarachnoid space and the epidural catheter was normally placed in the epidural space followed by injecting local anesthetics into the epidural space via the epidural catheter, where the dural puncture created a conduit for translocation of local anesthetics from the epidural space to the subarachnoid space which was a unique feature of DPE technique.

Our study assessed the efficacy of DPE with pencil point spinal needle (25-27 G) during elective CS. Primary outcome was the onset time of surgical anesthesia which is defined as the time from the end of the initial dose injection to when the bilateral sensory block level reached the T6 dermatome. secondary outcomes were number of patients with cranial sensory block toT6 Level, number of patients with a modified bromage score reaching 3 at 15 min, intraoperative IV analgesia, local anesthetic volume, incidence of vasopressor administration and maternal &fetal complications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (ASAI&II) with singleton vertex presentation cephalic presentation foetus at 38 to 42 weeksꞌ gestation.
* Age: 20-35 years old.
* Weight: 57-85 Kg.
* Height: 155-170cm.

Exclusion criteria

* Non-elective CS.
* Known foetal anomalies.
* Patient refusal or uncooperative patients.
* Patients with history of drug abuse and maternal diseases (i.e. diabetes mellitus, cardiac disease, heart block/dysrhythmia, hypertension, chronic obstructive respiratory disease, preeclampsia, eclampsia, placenta previa, placental abruption, coagulation abnormalities or hematological diseases).
* Spinal deformities, previous spinal surgeries, allergy to amide type of local anesthetics, localized skin sepsis at spinal lumbar region, neurological diseases, peripheral neuropathy, neuromuscular diseases, psychiatric diseases, hepatic and renal diseases, metabolic and endocrinal diseases and Raynaud's disease.
* Severe hypovolemia, severe hemodynamic instability and patients with anemia (Hb <10 gm %).
* Morbidly obese (BMI > 35 kg/m2) patients.
* Those who are very short (<150cm) or very tall (>170 cm).
* Patients on therapy with adrenergic receptor antagonist, anticoagulants, calcium channel blocker, and/or ACE inhibitor.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
was the onset time to surgical anesthesia | up to 20 minutes after local anesthetic injection
  was defined as the time from the end of the intraoperative epidural test dose injection [the start of epidural extension anaesthesia (time zero on the stopwatch)] to when the sensory block level reached the T6 dermatome bilaterally (when the patient could no longer feel sharp sensation at T6) (assessed bilaterally at the midclavicular line)

CONTACTS AND LOCATIONS:
Locations (1):
- Reham Ali Abdelhaleem Abdelrahman, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No